CLINICAL TRIAL: NCT00989066
Title: Brazil Xience V Everolimus-Eluting Coronary Stent System "Real-World" Outcomes Registry
Acronym: BRAVO
Status: Completed | Type: Observational
Sponsor: Cardiovascular Research Center, Brazil (Other)
Responsible Party: Sponsor
Other Study IDs: BRA01
Record Dates: First submitted 2009-10-01; First posted 2009-10-02 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-11

CONDITIONS: Arterial Coronary Disease
Keywords: Xience V; stent; coronary disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To evaluate the performance and long-term clinical outcomes of the Xience V everolimus-eluting coronary stent system (EECSS) in the treatment of minimally selective, high risk patients in the real-world clinical practice.

DETAILED DESCRIPTION:
Prospective, multicenter, non-randomized, post-marketing web-based registry.Patients all comers assigned for percutaneous coronary intervention (PCI) who present with at least one angiographically documented coronary artery lesion suitable for percutaneous treatment with implantation of Xience V EECSS only can be included on this Registry.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years of age; clinical indication for elective or emergency PCI with stent implantation of at least one angiographically documented coronary artery lesion; agreement to undergo ALL study protocol follow-ups
* Diseased coronary vessel(s) with the presence of at least one obstruction >50% diameter stenosis by visual estimation in a major epicardial vessel or a major branch (≥2.50mm), with anatomy suitable for percutaneous treatment with implantation of the Xience V EECSS

Exclusion Criteria:

* Known illness with life expectancy <24 months; impossibility to comply with all protocol follow-ups
* Coronary anatomy unsuitable for percutaneous treatment with implantation of the Xience V EECSS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients all comers assigned for percutaneous coronary intervention who present with at least one angiographically documented coronary artery lesion suitable for percutaneous treatment with implantation of Xience V
Sampling Method: Non-Probability Sample
Enrollment: 535 (Actual)
Dates: Start 2008-09; Primary Completion 2011-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Major Adverse Cardiac Events (MACE) at 12 months clinical follow-up | 12 months

SECONDARY OUTCOMES:
Rates of procedural success | 24 months
MACE at in-hospital | 30 days, 6 months, and 24 months
Toll-like receptor (TLR) | at 6 and 12 months
Stent thrombosis up to 24 mo | up to 24 months
Dual anti-platelet therapy compliance | at 1, 6 and 12 months
Major bleeding events | at 1, 6 and 12 mo

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Abizaid, MD, PhD, Principal Investigator — Cardiovascular Research Center
Locations (24):
- Brazil (24):
  - CIAS Unimed Vitória, Vitória, Espírito Santo
  - Encore, Goiânia, Goiás
  - Hospital Lifecenter, Belo Horizonte, Minas Gerais
  - Hospital Mater Dei, Belo Horizonte, Minas Gerais
  - Hospital Madre Tereza, Nova Lima, Minas Gerais
  - Instituto do Coração do Triângulo Mineiro, Uberlândia, Minas Gerais
  - Hospital Cardiológico Costantini, Curitiba, Paraná
  - Instituto de Neurologia de Curitiba, Curitiba, Paraná
  - Centro Interado de Medicina Intervencionista, Belém, Pará
  - Maximagem, Recife, Pernambuco
  - Hemocor, Jacarepaguá, Rio de Janeiro
  - Barra DOr, Rio de Janeiro, Rio de Janeiro
  - Hospital Copa DOr, Rio de Janeiro, Rio de Janeiro
  - Hospital Quinta DOr, Rio de Janeiro, Rio de Janeiro
  - Hospital São Vicente de Paulo, Passo Fundo, Rio Grande do Sul
  - Fundação Universitária de Cardiologia, Porto Alegre, Rio Grande do Sul
  - Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - Hospital São Lucas da PUC, Porto Alegre, Rio Grande do Sul
  - Santa Casa de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Albert Einstein, São Paulo, São Paulo
  - Hospital Bandeirantes, São Paulo, São Paulo
  - Hospital Beneficência Portuguesa, São Paulo, São Paulo
  - Hospital do Coração, São Paulo, São Paulo
  - Instituto Dante Pazzanese de Cardiologia, São Paulo, São Paulo